CLINICAL TRIAL: NCT03870659
Title: Value of Abbreviated Breast MRI in Cancer Detection
Brief Title: Abbreviated Breast MRI in Cancer Detection
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, AShassan, Principle investigator, Assiut University
Other Study IDs: Abbreviated Breast MRI
Record Dates: First submitted 2019-03-08; First posted 2019-03-12 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Breast MRI — Magnetic resonance imaging to the breast

SUMMARY:
Breast cancer is one of the leading causes of death among women, with early detection being the key to improve prognosis and survival.

Randomized controlled trials have found that screening mammography has decreased the mortality of breast cancer by 30%.

However, with a sensitivity of 70%, mammography has its limitations particularly in women with dense breasts.

The use of breast MRI for screening has increased over the past decade. Most experiences exist in women at elevated familial risk of breast cancer. In these women, MRI screening shifts the stage distribution of breast cancers toward lower stages and reduces the fraction of interval cancers.

Kuhl et al in 2014 were the first to report on the feasibility of an abbreviated breast MRI protocol for breast cancer screening. Their protocol consisting of an unenhanced T1-weighted and first contrast-enhanced T1-weighted sequence, subtraction imaging, and a single MIP image.

This groundbreaking study found that image acquisition and interpretation time could be reduced without having a negative impact on diagnostic accuracy.

DETAILED DESCRIPTION:
Breast MRI screening is associated with high direct and indirect costs. These, together with the lack of sites that offer high-level breast MRI, limit clinical access to screening MRIs.

One reason for the high cost is that current breast MRI protocols are time consuming to acquire and read. A typical MRI study occupies the MRI system for up to 40 minutes and generates several hundred images.

DCE-MRI allows the assessment of high-resolution breast morphology and enhancement kinetics to depict angiogenesis as a tumor-specific feature. At any given field strength, DCE-MRI is the most sensitive modality for breast cancer detection, with a pooled sensitivity of 93%; DCE-MRI has good pooled specificity of 71%.

With the abbreviated MRI protocol, the acquisition time was substantially decreased to 3 minutes, compared with 17 minutes for the full diagnostic protocol. The interpretation time of the abbreviated protocol was 28 seconds on average and 2.8 seconds when the MIP image alone was evaluated.

ELIGIBILITY:
Inclusion Criteria:

- All women referred to our radiology department at assiut university hospital for performing breast MRI

Exclusion Crieria:

* no exclusion criteria

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Women referred for performing breast MRI to exclude presence of breast cancer and their lesion characterization
Sampling Method: Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
To evaluate accuracy of abbreviated breast MRI in cancer detection | 2 years
  Sensitivity and specificity of abbreviated breast MRI in detection of cancer will be calculated and compared to those of the full protocol

CONTACTS AND LOCATIONS:
Overall Officials: Abeer, PhD, Study Director — Assiut University
Locations (1):
- Zahraa, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided